CLINICAL TRIAL: NCT06740591
Title: Evaluation of the Efficacy and Safety of High-Definition Transcranial Direct Current Stimulation for Pain Reduction in Post-Stroke Pain Patients: Investigator-Initiated, Single-Center, Randomized, Crossover, Single-Blind Clinical Trial
Brief Title: HD-tDCS for Pain Reduction in Post-Stroke Pain: a Randomized Crossover Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 23-2023-001
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Pain; CPSP; TDCS
MeSH Terms: conditions — Stroke; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental : HD-tDCS (Experimental): The HD-tDCS stimulation was applied for 20 minutes, 5 times a week, over a total of 10 sessions.
  Interventions: Device: HD-tDCS
- Sham HD-tDCS (Sham Comparator): The Sham HD-tDCS stimulation was applied for 20 minutes, 5 times a week, over a total of 10 sessions.
  Interventions: Device: Sham High-Definition Transcranial Direct Current Stimulation(sham HD-tDCS)

INTERVENTIONS:
Device: HD-tDCS — The HD-tDCS stimulation was applied for 20 minutes, 5 times a week, for a total of 10 sessions.
  Arms: Experimental : HD-tDCS
Device: Sham High-Definition Transcranial Direct Current Stimulation(sham HD-tDCS) — The Sham HD-tDCS stimulation was applied for 20 minutes, 5 times a week, for a total of 10 sessions.
  Arms: Sham HD-tDCS

SUMMARY:
This study aims to assess the effectiveness of multichannel transcranial direct current stimulation (tDCS) in alleviating pain and to evaluate its safety in patients with central post-stroke pain (CPSP)

ELIGIBILITY:
Inclusion Criteria :

* Adults aged between 19 and 90 years.
* Diagnosed with first-ever stroke based on clinical observation and neuroimaging by a physician.
* Stroke lesion located in the cortex or subcortex [basal ganglia (BG) or thalamus].
* Fulfillment of mandatory criteria for pain (pain in the body part corresponding to central nervous system lesions, onset of pain immediately after stroke, confirmation that the pain corresponds to the lesion site, exclusion of other causes of pain such as peripheral neuropathic pain).
* Cognitive ability sufficient to understand and follow the instructions of the researcher.
* Voluntary consent to participate in the clinical trial and signed informed consent.

Exclusion Criteria :

* History of fractures or orthopedic surgeries on the affected side.
* Presence of significant pre-existing neurogenic disorders.
* Co-existing severe psychiatric disorders such as major depressive disorder, schizophrenia, bipolar disorder, or dementia.
* Complex regional pain syndrome (CRPS) diagnosed based on Budapest criteria.
* Other causes of pain in the affected area, such as peripheral nerve damage.
* Exclusion criteria for transcranial magnetic stimulation (e.g., pregnancy, cancer, patients with abnormal responses to stimulation, presence of intracranial metal implants, hypersensitivity to pain, history of seizures, or injuries/skin conditions at electrode attachment sites).
* Deemed unsuitable for participation in the study by the principal investigator.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Change of pain score in Brief Pain Inventory(BPI) | Baseline(prior to the first intervention), Week 2(after the end of the first device intervention), Week 3(prior to the second device intervention), and Week 4(after the end of the second device intervention)
  The Brief Pain Inventory (BPI) is a widely used questionnaire for assessing pain. It measures pain intensity over the past week or the last 24 hours using four 11-point Likert scale items: worst pain, least pain, average pain, and current pain. Additionally, it evaluates how pain interferes with daily activities, mood, walking ability, normal work, relationships with others, sleep, and leisure activities, also using an 11-point Likert scale. The total score ranges from 0 (no pain) to 40 (worst pain), with higher scores indicating greater musculoskeletal pain severity. Pain intensity is categorized as mild (1-4), moderate (5-6), or severe (7-10).

SECONDARY OUTCOMES:
Change of pain score in Neuropathic Pain Scale(NPS) | Baseline(prior to the first intervention), Week 2(after the end of the first device intervention), Week 3(prior to the second device intervention), and Week 4(after the end of the second device intervention)
  The Neuropathic Pain Scale (NPS) consists of 10 subscales, each representing a different aspect of neuropathic pain. Pain intensity for each subscale is measured using a Visual Analog Scale (VAS), where 0 indicates no pain and 10 represents the worst possible pain. These subscales assess the intensity of overall pain, sharpness, heat, aching, cold, sensitivity to light touch or fabric, and itchiness. Participants complete this assessment through an interview-based questionnaire. Higher scores reflect greater pain intensity.
Change of depression score in Beck Depression Inventory-II(BDI-II) | Baseline(prior to the first intervention), Week 2(after the end of the first device intervention), Week 3(prior to the second device intervention), and Week 4(after the end of the second device intervention)
  The Beck Depression Inventory (BDI) is one of the most widely used depression assessment tools worldwide. The BDI consists of questions based on common daily life experiences . As a self-report tool, participants complete the questionnaire by indicating which statements apply to them. The inventory includes 21 items, each with four response options, scored from 0 to 3, with a total possible score of 63. Higher scores indicate a greater severity of depression.
Change of quality of life score in the EuroQol Five-dimensions-Three-Level Quality of Life Instrument(EQ-5D-3L) | Baseline(prior to the first intervention), Week 2(after the end of the first device intervention), Week 3(prior to the second device intervention), and Week 4(after the end of the second device intervention)
  This tool is widely used to assess health-related quality of life. It consists of three multiple-choice questions across five domains: mobility (M), self-care (SC), usual activities (UA), pain/discomfort (PD), and anxiety/depression (AD). Responses are coded on a scale from 1 to 3, representing none, moderate, and severe, respectively. The total score ranges from 1 (no problems in any domain) to 3 (severe problems in all domains). Higher scores indicate a lower quality of life.
Change in Blood Pressure to Sustained Muscle Contraction | Baseline(prior to the first intervention), Week 2(after the end of the first device intervention), Week 3(prior to the second device intervention), and Week 4(after the end of the second device intervention)
  This assessment evaluates the autonomic nervous system's response to sustained muscle contraction by measuring blood pressure. Blood pressure are measured while the participant is lying comfortably for 20 minutes in a relaxed state. Then, the participant holds a hand dynamometer at 30% of their maximum grip strength for 5 minutes, during which blood pressure are recorded. Afterward, the participant rests for 10 minutes in a relaxed position, and the measurements are taken again.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Il Shin, Dr., Study Director — Pusan National University Yangsan Hospital
Locations (1):
- Pusan national university Yangsan Hospital, Gyeongsang, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No